CLINICAL TRIAL: NCT07392671
Title: Investigation of the Effects of Limbic System-Oriented Combined Manual Therapy on Pain, Joint Range of Motion, Muscle Strength, Joint Position Sense, Balance, Functional Status, Emotional State, Quality of Life, and Sleep Quality in Temporomandibular Joint Dysfunction
Brief Title: Investigation of the Effects of Different Treatment Approaches in Jaw (Temporomandibular) Joint Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Polen Hazımoğlu, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-22078
Record Dates: First submitted 2026-01-12; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Disorders (TMDs)
Keywords: temporomandibular joint disorders; Physiotherapy; Manual therapy; Limbic system; Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: This study was designed as a parallel-group interventional clinical trial. Participants who agreed to participate in the study were randomly assigned into two groups using a block randomization method. Each group received a different physiotherapy and rehabilitation program during the same study period. Recruitment has been completed, and no new participants are being enrolled. Participants continue to receive the assigned interventions and complete the planned assessments while remaining in their allocated groups throughout the study.
Who Masked: Participant
Masking Description: Only participants were blinded to group allocation. No other parties were masked in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Manual Therapy + Exercise Program (Active Comparator): Participants in this arm receive a conventional physiotherapy and rehabilitation program consisting of manual therapy applied to the temporomandibular joint and cervical region, supervised therapeutic exercises, and a structured home exercise program. No limbic-oriented manual therapy techniques are included in this arm.
  Interventions: Other: Conventional Physiotherapy and Rehabilitation Program
- Conventional Program + Limbic-Oriented Manual Therapy (Experimental): Participants in this arm receive the same conventional physiotherapy and rehabilitation program, including temporomandibular joint and cervical manual therapy, supervised therapeutic exercises, and a home exercise program, with the addition of limbic-oriented manual therapy techniques aimed at modulating central pain processing and emotional regulation.
  Interventions: Other: Conventional Physiotherapy and Rehabilitation Program; Other: Limbic-Oriented Manual Therapy

INTERVENTIONS:
Other: Conventional Physiotherapy and Rehabilitation Program — The intervention is delivered over a 6-week period. Manual therapy techniques applied to the cervical region and temporomandibular joint, along with supervised jaw exercises, are administered twice per week. In addition, participants perform postural exercises as part of a home exercise program for 6 weeks, 5 days per week, three times per day, with 10 repetitions per exercise. All interventions are administered by a physiotherapist according to a standardized physiotherapy protocol.
Other: Limbic-Oriented Manual Therapy — In addition to the conventional physiotherapy and rehabilitation program, limbic-oriented manual therapy techniques are applied over a 6-week period. Three limbic-oriented manual therapy techniques are administered during each session, with each technique applied for an average duration of approximately 3 minutes. These techniques are administered twice per week by a physiotherapist according to the study protocol. The limbic-oriented manual therapy is delivered alongside manual therapy to the cervical region and temporomandibular joint, supervised jaw exercises, and a structured home exercise program.
  Arms: Conventional Program + Limbic-Oriented Manual Therapy

SUMMARY:
Temporomandibular joint disorders (TMD) are common conditions that may cause jaw pain, limited jaw movement, and reduced quality of life. Individuals with TMD can also experience neck-related problems, balance impairments, emotional changes, and sleep disturbances.

This interventional study aims to investigate the effects of a combined physiotherapy and rehabilitation program in individuals with temporomandibular joint dysfunction. The intervention consists of conventional manual therapy techniques applied to the temporomandibular joint and cervical region, combined with specific manual therapy techniques targeting the limbic system, along with therapeutic exercise applications.

The study will evaluate the effects of this combined treatment approach on pain, jaw range of motion, joint position sense, balance, emotional status, patient satisfaction, and quality of life and sleep in individuals with TMD.

DETAILED DESCRIPTION:
Temporomandibular joint dysfunction is a complex condition that affects the masticatory system and is frequently associated with cervical musculoskeletal impairments, altered sensorimotor control, and psychosocial factors. In addition to local biomechanical dysfunctions, individuals with temporomandibular disorders may experience changes in pain processing, emotional regulation, balance, and overall quality of life. These factors highlight the need for a comprehensive rehabilitation approach that addresses both peripheral and central mechanisms.

Physiotherapy and rehabilitation interventions for temporomandibular joint dysfunction traditionally focus on the temporomandibular joint and cervical region using manual therapy techniques and therapeutic exercises. While these approaches are effective in improving physical impairments, emerging evidence suggests that central mechanisms, including the limbic system, may influence pain perception, emotional status, and functional outcomes in individuals with temporomandibular disorders.

This interventional study is designed to investigate the effects of a combined physiotherapy and rehabilitation approach that integrates conventional manual therapy techniques applied to the temporomandibular joint and cervical region with specific manual therapy techniques oriented toward the limbic system, along with therapeutic exercise applications. The combined approach aims to address musculoskeletal, sensorimotor, and emotional components of temporomandibular joint dysfunction within a holistic rehabilitation framework.

Participants diagnosed with temporomandibular joint dysfunction will undergo the intervention program and will be evaluated before and after the treatment period. The study focuses on changes in pain, jaw function, sensorimotor control, balance, emotional status, patient satisfaction, and quality of life and sleep, providing a multidimensional assessment of treatment effects.

By examining the outcomes of this combined intervention, the study seeks to enhance the understanding of integrative physiotherapy strategies in the management of temporomandibular joint dysfunction and to support the development of more comprehensive rehabilitation approaches that consider both physical and emotional aspects of the condition.

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 and 60 years

Diagnosed with temporomandibular joint dysfunction (TMD - disc displacement or degenerative joint disease) by an Oral and Maxillofacial Surgery specialist

Clinical findings consistent with temporomandibular joint dysfunction

Presence of symptoms and pain related to TMD for at least 6 months

No history of acute trauma, infection, or neurological disease

No limitation of joint range of motion in the angles assessed for joint position sense

No history of any treatment or physiotherapy for TMD within the last 6 months

Not using occlusal splints, orthodontic appliances, and/or medications for pain

Use of no more than one fixed prosthetic restoration (bridge or implant-supported crown) in a single region

Voluntary participation and provision of written informed consent

Exclusion Criteria:

History of jaw and/or cervical region surgery or trauma within the last 6 months

Presence of rheumatological or psychiatric disorders

History of fracture involving the temporomandibular joint, cervical, or upper thoracic region

Presence of acute cervical disc pathology or other acute conditions affecting the cervical region

Presence of skin infection or open wounds

Presence of perceptual or communication disorders

Partial edentulism classified as Kennedy Class I, II, or III, or multiple missing teeth that impair masticatory function, except for single-tooth loss

Presence of fixed prosthetic restorations for more than one missing tooth

Use of removable partial or complete dentures

Unwillingness to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity at Rest (Visual Analog Scale) | Baseline and after 6 weeks
  Pain intensity at rest is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates no pain and a score of 10 indicates the worst imaginable pain.
  Higher scores represent greater pain intensity. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Pressure Pain Threshold (Algometry) | Baseline and after 6 weeks
  Pressure pain threshold is assessed using a handheld pressure algometer. Measurements are performed bilaterally at three anatomical sites: the temporomandibular joint region, masseter muscle, and temporalis muscles, and recorded in Newton (N).
  At each site, three consecutive measurements are taken, and the mean value is calculated for analysis.
  Higher values indicate greater pressure pain tolerance, whereas lower values indicate increased pain sensitivity.
  Assessments are conducted at baseline and at the end of the treatment period.
Cervical Joint Position Sense | Baseline and after 6 weeks
  Cervical joint position sense is assessed during flexion-extension, right and left rotation, and right and left lateral flexion movements using target angle tests and the head repositioning test. Flexion, extension, and rotation movements are assessed at mid-range positions (50% of the available range of motion) and at target angles of 10° and 30°. Lateral flexion movements are assessed at target angles of 10° and 20°, as well as at mid-range positions (50% of the available range of motion). During each test, the deviation from the target angle is recorded. The angular error is calculated as the absolute difference between the target angle and the angle achieved by the participant and recorded in degrees (°). Higher angular error values indicate poorer joint position sense, whereas lower values indicate better proprioceptive accuracy. Each test is performed three times with the participant's eyes closed, and the mean value of the three measurements is recorded for analysis.
Temporomandibular Joint Range of Motion | Baseline and after 6 weeks
  Temporomandibular joint range of motion is assessed using a digital caliper. Pain-free maximum mouth opening, right and left lateral excursions, and mandibular protrusion movements are measured.
  All measurements are recorded in millimeters (mm) for analysis. Higher values indicate greater mandibular mobility, whereas lower values indicate restricted temporomandibular joint range of motion.
Cervical Joint Range of Motion | Baseline and after 6 weeks
  Cervical joint flexion, extension, bilateral lateral flexion, and rotation movements are evaluated using a cervical range of motion (CROM) device.
  Measurements are recorded in degrees (°). Higher values indicate greater cervical mobility, whereas lower values indicate restricted cervical range of motion.
Static Balance (Flamingo Balance Test) | Baseline and after 6 weeks
  Static balance is assessed using the Flamingo Balance Test. Participants are instructed to stand on a wooden balance beam and maintain balance on one lower extremity.
  The test is performed on the participant's dominant extremity. Timing begins when the participant achieves single-leg stance, and the participant is asked to maintain balance for one minute without falling.
  During the one-minute period, each attempt to regain balance after a loss of balance is counted.
  The total number of balance attempts recorded during the test constitutes the participant's score.
  Higher scores indicate poorer static balance performance, whereas lower scores indicate better balance control.
Dynamic Balance (Y Balance Test) | Baseline and after 6 weeks
  Dynamic balance is assessed using the Y Balance Test. The test is performed in the anterior, posteromedial, and posterolateral directions.
  Participants perform three trials in each direction, and the mean value of the three measurements is calculated for analysis.
  Reach distances are recorded in centimeters (cm). Higher reach distances indicate better dynamic balance performance, whereas lower values indicate reduced balance ability.
Pain Intensity During Chewing (Visual Analog Scale) | Baseline and after 6 weeks
  Pain intensity during chewing is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  Pain is evaluated separately during chewing of hard and soft food. A score of 0 indicates no pain, and a score of 10 indicates the worst imaginable pain.
  Higher scores represent greater pain intensity. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Pain Intensity During Biting (Visual Analog Scale) | Baseline and after 6 weeks
  Pain intensity during biting is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates no pain, and a score of 10 indicates the worst imaginable pain.
  Higher scores represent greater pain intensity. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Pain Intensity During Night-Time (Visual Analog Scale) | Baseline and after 6 weeks
  Night-time pain intensity is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates no pain, and a score of 10 indicates the worst imaginable pain.
  Higher scores represent greater pain intensity. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Pain Intensity During Yawning | Baseline and after 6 weeks
  Pain intensity during yawning is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates no pain, and a score of 10 indicates the worst imaginable pain.
  Higher scores represent greater pain intensity. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Pain Intensity During Eating (Visual Analog Scale) | Baseline and after 6 weeks
  Pain intensity during eating is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates no pain, and a score of 10 indicates the worst imaginable pain.
  Higher scores represent greater pain intensity. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Temporomandibular Joint Dysfunction Severity (Fonseca Anamnestic Questionnaire) | Baseline and after 6 weeks
  Temporomandibular joint functional status is assessed using the Turkish version of the Fonseca Anamnestic Questionnaire. The total score ranges from 0 to 100, with higher scores indicating greater severity of temporomandibular joint dysfunction.
Mandibular Functional Impairment (Mandibular Function Impairment Questionnaire) | Baseline and after 6 weeks
  Mandibular functional status is assessed using the Turkish version of the Mandibular Function Impairment Questionnaire. The total score ranges from 0 to 68, with higher scores indicating greater functional impairment

SECONDARY OUTCOMES:
Chewing Quality (Visual Analog Scale) | Baseline and after 6 weeks
  Chewing quality is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates very poor chewing quality, and a score of 10 indicates excellent chewing quality.
  Higher scores represent better chewing quality. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Patient Satisfaction With Treatment (Visual Analog Scale) | At the end of the treatment period (6 weeks)
  Patient satisfaction with the treatment is assessed using the Visual Analog Scale (VAS), a 10-cm horizontal line ranging from 0 to 10 cm.
  A score of 0 indicates "not satisfied at all," and a score of 10 indicates "extremely satisfied." Higher scores represent greater treatment satisfaction. The distance from the left end of the scale to the marked point is measured using a ruler and recorded in centimeters (cm).
Postural Assessment | Baseline and after 6 weeks
  Postural assessment is performed bilaterally using a measuring tape. Linear distances are measured between predefined anatomical landmarks and recorded in centimeters (cm). Measurements are obtained from both sides of the body for analysis.
Deep Cervical Flexor Muscle Strength | Baseline and after 6 weeks
  Deep cervical flexor muscle strength is assessed using a Stabilizer Pressure Biofeedback unit.
  The pressure generated by the participant during the test is recorded in millimeters of mercury (mmHg).
  The assessment is performed under two conditions: without visual feedback and with visual feedback, during which the manometer is visible to the participant.
  In both conditions, participants are instructed to perform a craniocervical flexion movement, and the corresponding pressure values are recorded for analysis.
  Higher pressure values indicate greater deep cervical flexor muscle activation and strength.
Neck Disability | Baseline and after 6 weeks
  Neck-related disability is assessed using the Turkish version of the Neck Disability Index (NDI) questionnaire.
  The total score ranges from 0 to 50, with higher scores indicating greater neck-related disability and functional limitation.
Health-Related Quality of Life (WHOQOL-BREF) | Baseline and after 6 weeks
  QQuality of life is assessed using the Turkish validated version of the World Health Organization Quality of Life Questionnaire-Brief Form (WHOQOL-BREF). Domain scores are transformed to a 0-100 scale, with higher scores on the questionnaire indicating better perceived quality of life.
Sleep Quality (Pittsburgh Sleep Quality Index) | Baseline and after 6 weeks
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Emotional Status - Depression (Beck Depression Inventory) | Baseline and after 6 weeks
  Emotional status related to depressive symptoms is assessed using the Beck Depression Inventory (BDI). The total score ranges from 0 to 63, with higher scores indicating greater severity of depressive symptoms.
Emotional Status - Anxiety (Beck Anxiety Inventory) | Baseline and after 6 weeks
  Emotional status related to anxiety symptoms is assessed using the Beck Anxiety Inventory (BAI). The total score ranges from 0 to 63, with higher scores indicating greater severity of anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Musculoskeletal Physiotherapy and Rehabilitation Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the research team. The data are collected as part of a doctoral thesis and will be used only for the purposes defined in the study protocol and related scientific publications, in accordance with ethical approval and data protection regulations.